CLINICAL TRIAL: NCT04638634
Title: A Single Center, Phase 1, Single-Ascending Dose, Open-Label Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of CSL760, an Intravenous Anti-SARS-CoV-2 Hyperimmune Globulin, in Healthy Adult Subjects
Brief Title: Pharmacokinetics, Safety, and Tolerability of CSL760, an Intravenous Anti-SARS-CoV-2 Hyperimmune Globulin, in Healthy Adult Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: For business reasons, not a safety issue
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CSL760_1001
Record Dates: First submitted 2020-11-19; First posted 2020-11-20 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Coronavirus Disease 2019 (COVID-19)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSL760 (low dose) (Experimental): Administered as an intravenous infusion
  Interventions: Biological: CSL760
- CSL760 (high dose) (Experimental): Administered as an intravenous infusion
  Interventions: Biological: CSL760

INTERVENTIONS:
Biological: CSL760 — An Intravenous Anti-SARS-CoV-2 Hyperimmune Globulin
  Other Names: COVID-19 Immunoglobulin-VF

SUMMARY:
CSL760 is a human hyperimmune product of the purified gamma immunoglobulin (IgG) fraction of human plasma containing polyvalent neutralizing antibodies to SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2). CSL is evaluating CSL760 as a passive immunotherapy for COVID-19 (Coronavirus Disease 2019).

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 65 years of age
* Female subjects must be postmenopausal or have a negative pregnancy test
* Body weight in the range of ≥ 50 kg and ≤ 100 kg and have a body mass index of ≥ 18 to ≤ 32 kg/m2

Exclusion Criteria:

* History of acute or chronic renal failure, thromboembolism, chronic respiratory illness, aseptic meningitis syndrome, or recurrent severe headaches or migraines.
* Positive viral serology test for HIV -1/2 antibody, hepatitis B virus surface antigen, or hepatitis C virus antibody
* Positive viral serology test for SARS-CoV-2 antibodies
* Received any live viral or bacterial vaccinations within 8 weeks
* Evidence of current active infection.
* Known malignancy or a history of malignancy in the past 5 years
* Female subject of childbearing potential or fertile male subject either not using or not willing to use an acceptable double barrier method of contraception to avoid pregnancy during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Total immunoglobulin (IgG) concentration of CSL760 | At 0,0.5,1,2,6,12,24, and 48 hours, and 7,14,28,49, and 91 days after end of IV infusion
Maximum concentration (Cmax) of CSL760 | Up to 91 days after end of IV infusion
Time of Cmax (tmax) of CSL760 | Up to 91 days after end of IV infusion
Area under the concentration-time curve (AUC) from time 0 to the last measurable concentration (AUC0-last) of CSL760 | Up to 91 days after end of IV infusion

SECONDARY OUTCOMES:
Number of subjects with Treatment-emergent adverse events (TEAEs) | From start of infusion up to 91 days
Percent of subjects with TEAEs | From start of infusion up to 91 days
Number of subjects with Serious adverse events (SAEs) | From start of infusion up to 91 days
Percent of subjects with SAEs | From start of infusion up to 91 days
Number of subjects with Clinically significant laboratory abnormalities that are reported as adverse events (AEs) | From start of infusion up to 91 days
Percent of subjects with Clinically significant laboratory abnormalities that are reported as AEs | From start of infusion up to 91 days

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Innovation Pty Ltd
Locations (1):
- CMAX Clinical Research, Adelaide, Australia

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider requests to share Individual Patient Data (IPD) from systematic review groups or bona-fide researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.
Supporting Information: Study Protocol, SAP
Time Frame: IPD requests may be submitted to CSL no earlier than 12 months after publication of the results of this study via an article made available on a public website.
Access Criteria: Requests may only be made by systematic review groups or bona-fide researchers whose proposed use of the IPD is non-commercial in nature and has been approved by an internal review committee.
  An IPD request will not be considered by CSL unless the proposed research question seeks to answer a significant and unknown medical science or patient care question as determined by CSL's internal review committee.
  The requesting party must execute an appropriate data sharing agreement before IPD will be made available.